CLINICAL TRIAL: NCT05812300
Title: The Clinical Study of Injection of Freshly Prepared HA35 for Treatment Gingivitis
Brief Title: Local Injection of Periodontal Pocket Method for the Treatment of Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSHN003
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HA35 local injection of Periodontal Pocket group (Experimental): The tissue-permeable 35 kDa low molecular hyaluronan fragment HA35 was freshly manufactured using pharmaceutical grade hyaluronidase PH20 injection (State Drug Administration H31022111) and joint cavity HA injection (State Drug Administration H20174089) mixed at room temperature for 20 min.
  Interventions: Drug: Freshly manufactured 35 kDa hyaluronan fragment

INTERVENTIONS:
Drug: Freshly manufactured 35 kDa hyaluronan fragment — The study was an open-label clinical trial. A pre- and posttreatment controlled study approach was used, whereby the investigator injected 35 kDa hyaluronan fragment HA35 into the periodontal pocket in a single dose of 100 mg. The distribution of the injection amount was determined by the location of gingival inflammation.
  Other Names: HA35

SUMMARY:
Preliminary clinical studies have confirmed that injection of freshly prepared HA35 can reduce symptoms and signs of gingivitis or periodontitis. This clinical study is a prospective repeated experiments. The purpose of this study was to verify the effectiveness of HA35 injection therapy.

DETAILED DESCRIPTION:
The previous studies showed that toothpastes containing the cosmetic grade raw material of the 35 kDa low molecular hyaluronan fragment HA35 significantly reduced symptoms and signs of gingivitis or periodontitis. In this study, patients with mild to moderate periodontitis suffering from symptoms and signs, including discomfort and swelling and bleeding of periodontal tissue, were treated by intrapocket injection of freshly manufactured hyaluronan fragment HA35. This study is an repeat clinical study comparing pre- and posttreatment effects similar to others.

ELIGIBILITY:
Inclusion Criteria:

* Healthy condition and with a clinical diagnosis of mild to moderate gingivitis.
* Male or female volunteers aged 18-60 years.
* Gingival Index (GI) from 1 to 2 (0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing)

Exclusion Criteria:

* Healthy condition and with a clinical diagnosis of severe gingivitis.
* Pregnant or lactating females.
* Be concomitantly participating in another clinical study.
* History of any allergic reaction to HA.
* To treat the gingivitis with any other medication/mouthwashes in the period of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Measurement of gum discomfort | 7 days
  Each patient rated their gingival discomfort or itching on a scale of 0 to 10. 0 means "no", and 10 means "the most".
Measurement of gum redness and swelling | 7 days
  The physician used the numbers 0-10 to rate the intensity of gingival redness and swelling in the subject. 0 means "no"; 10 means "highest".
Measurement of probe gingival bleeding | 7 days
  The physician used the numbers 0-10 to rate the extent to which the subject's probe gums were bleeding. A score of 0 indicated "no" and 10 indicated "the most"

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: No
The data will be sent to the accepting journal study.